CLINICAL TRIAL: NCT00275743
Title: Dynamic MRI - A Novel Approach for Measuring Gastric Accommodation
Brief Title: Use of MRI for Assessing Stomach Relaxation in Response to a Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Adil Bharucha, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-004022
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Dyspepsia; Healthy Volunteers
MeSH Terms: conditions — Dyspepsia

INTERVENTIONS:
Procedure: MRI

SUMMARY:
This study is being done to test new way of measuring the relaxation of the stomach after a meal (called gastric accommodation) by using a MRI scan. This new test will be compared with the standard test of measuring stomach relaxation that uses radioactive tracers. These tests will be compared in healthy volunteers and people with upper abdominal symptoms (known as dyspepsia).

ELIGIBILITY:
Inclusion criteria for Dyspeptic patients (30 required)

* One or more of eight postprandial dyspeptic symptoms i.e. fullness, bloating, epigastric discomfort, early satiety, nausea, vomiting, belching, pain for a minimum of 3 months, OR
* Patients fulfilling the ROME-II criteria for functional dyspepsia,
* AND no symptom improvement after standard dose PPI treatment,
* AND normal upper gastrointestinal endoscopy within six months prior to the study

Inclusion Criteria for Healthy Controls (20 required)

• Absence of current abdominal symptoms or depression

Exclusion Criteria for all Participants

* Known structural upper GI disorder (e.g. peptic ulcer disease, esophagitis, malignancy);
* Abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, tubal ligation, or inguinal hernia repair;
* Medications that may alter gastrointestinal motility, e.g., serotoninergic agents, alpha adrenergic agonists, calcium channel or beta blockers; stable dose of thyroxine will be permitted;
* Pregnant or breast-feeding females;
* Known claustrophobia;
* Any metal objects in the body (e.g. metal implants, pacemaker, AICD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Gastric Volume (fasting and postprandial)
Antral Contractility

CONTACTS AND LOCATIONS:
Overall Officials: Adil E. Bharucha, M.B.B.S., M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States